CLINICAL TRIAL: NCT02816268
Title: Contact Force Guided Ablation Versus Conventional Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation
Acronym: FULL CONTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-DHM-21
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Improving Outcome After Pulmonary Vein Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Pulmonary vein isolation (Other): Conventional pulmonary vein isolation was gained by using an irrigated tip ablation catheter
  Interventions: Other: Pulmonary vein isolation
- Contact force pulmonary vein isolation (Other): Contact force was meassured by using the SMART-Touch ablation catheter (Biosense-Webster®)
  Interventions: Other: Pulmonary vein isolation

INTERVENTIONS:
Other: Pulmonary vein isolation

SUMMARY:
The investigators prospectively investigate the differences between contact-force guided pulmonary vein isolation (PVI) and conventional pulmonary vein isolation in patients with paroxysmal atrial fibrillation (PAF) with respect to adenosine guided unmasking of dormant conduction, procedural and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>=18 und < 80 years) with symptomatic paroxysmal AF
* At least one unsuccessful attempt of antiarrhythmic drug (betablocker or class I oder III).
* Oral anticoagulation with phenprocoumone, warfarine or DOAKs for at least 4 weeks prior to ablation with weekly documented INR > 2..
* Withdrawal of antiarrhythmic drugs at least 3 half times prior to ablation except amiodarone.

Exclusion Criteria:

* Left atrial thrombus
* Contraindications for oral anticoagulation or adenosin

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of reconnected pulmonary vein after ablation and a waíting period of 20min | 20min after procedure

SECONDARY OUTCOMES:
Time to first documented recurrence of atrial fibrillation | 12 month
Complications due to ablation | 30 days
Number of reconnected pulmonary veins | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes